CLINICAL TRIAL: NCT03479489
Title: A Prospective Case Series for Closed Hemorrhoidectomy - Efficacy of External Hemorrhoid Repair Using a Dehydrated Human Amnion Chorion Membrane
Brief Title: Use of Human Dehydrated Amnion Chorion Allograft in Closed Hemorroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFSUR001
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: External Hemorrhoid; External Hemorrhoid Thrombosed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human dehydrated amnion/chorion allofraft (Experimental): Closed hemorrhoidectomy patched with human dehydrated amnion chorion allograft
  Interventions: Other: Human dehydrated amnion chorion allograft

INTERVENTIONS:
Other: Human dehydrated amnion chorion allograft — Closed hemorrhoidectomy patched with dehydrated human amnion chorion allograft

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of human dehydrated amnion chorion allograft in closed hemorrhoidectomy as assessed by patient and wound assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of acutely thrombosed hemorrhoid or an external hemorrhoid exceeding 72 hours in duration
2. Subject is undergoing closed hemorrhoidectomy as their definitive treatment for the Grade 2-4 hemorrhoid
3. Subject is age 18 or older
4. Subject is willing and able to provide informed consent and participate in all procedures and follow-up evaluations necessary to complete the study

Exclusion Criteria:

1. Subject has a known history of poor compliance with medical treatments
2. Subject has signs and symptoms of active cirrhosis
3. Subject has signs and symptoms of Crohn's disease complicated by perianal manifestations
4. Subject is currently taking immunosuppressive medications
5. Subject has had previous surgery in the target area within the past 6 months prior to treatment or plans to have surgery other than closed hemorrhoidectomy in the target area within 180 days of treatment
6. Subject is currently receiving radiation therapy or chemotherapy
7. Subject has used an investigational drug, device or biologic within 12 weeks prior to treatment
8. Subject is pregnant at enrollment or is planning to become pregnant within 180 days of treatment; subject intends to breastfeed during the course of the trial
9. Subject has any significant medical condition(s) that, in the opinion of the Investigator, would interfere with protocol evaluation and participation
10. Subject has an allergy or known sensitivity to aminoglycoside antibiotics such as gentamicin sulfate and/or streptomycin sulfate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Reported Patient Pain | 60 days
  The primary endpoint of the study is the change in patient reported pain across four categories from baseline within the 60 day follow-up period. In every patient diary, subjects will be asked to assess their pain on a 10 point Likert scale under the following conditions
  * Do you experience pain continuously?
  * Do you experience pain with activity?
  * Do you experience pain while sitting?
  * Do you experience pain with bowel movements?

CONTACTS AND LOCATIONS:
Overall Officials: Donald Fetterolf, MD, Study Director — MiMedx Group, Inc.
Locations (1):
- Boulder Valley Surgical Associates, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No